CLINICAL TRIAL: NCT03062813
Title: The Therapy of Tacrolimus Combined With Entecavir on HBV Associated Glomerulonephritis : A Multicenter, Prospective, Randomized, Controlled, Single-blind Trial.
Brief Title: Tacrolimus Combined With Entecavir on HBV Associated Glomerulonephritis(HBV-GN)
Acronym: TOHBVGN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZMYe
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis B Virus Associated Nephrotic Syndrome
Keywords: Hepatitis B virus, tacrolimus,membranous nephropathy
MeSH Terms: conditions — Hepatitis B; Glomerulonephritis, Membranous | interventions — Tacrolimus; entecavir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus & entecavir (Experimental): Tacrolimus capsule, 0.5mg/capsule,1.0mg/capsule, 0.05-0.1mg/kg.d by mouth , every 12 hours for a day.Entecavir 0.5mg tablet by mouth every night.
  Interventions: Drug: Tacrolimus &entecavir
- placebo & entecavir (Active Comparator): Tacrolimus capsule, 0.5mg/capsule,1.0mg/capsule, 0.05-0.1mg/kg.d by mouth , every 12 hours for a day.Entecavir 0.5mg tablet by mouth every night.
  Interventions: Drug: placebo & entecavir

INTERVENTIONS:
Drug: Tacrolimus &entecavir — HBV-GN patients with nephrotic syndrome were randomly givenTacrolimus (0.05-0.1 mg/kg/day) combined with entecavir. Tacrolimus was divided into two daily doses at 12-hour intervals. Subsequent doses were adjusted to achieve a whole blood 12-hour trough level between 5 and 10 ng/ml.All patients will receive entecavir antiviral therapy(0.5mg/d), entecavir was taken once a day. All of HBV-GN patients were followed up to 25week.
  Other Names: FK506,Prograf, baraclude
  Arms: Tacrolimus & entecavir
Drug: placebo & entecavir — HBV-GN patients with nephrotic syndrome were randomly givenTacrolimus placebo (0.05-0.1 mg/kg/day) combined with entecavir.Tacrolimus placebo was divided into two daily doses at 12-hour intervals. All patients will receive entecavir antiviral therapy(0.5mg/d), entecavir was taken once a day. All of HBV-GN patients were followed up to 25week.
  Other Names: baraclude
  Arms: placebo & entecavir

SUMMARY:
This study was to evaluate the efficacy and safety of Tacrolimus combined with entecavir antiviral therapy for HBV-associated glomerulonephritis in china. Tacrolimus combined with entecavir rapidly and effectively induced remission of HBV-GN in Chinese adults. Meanwhile, Tacrolimus may have a synergistic antiviral effect with entecavir. The study protocol was reviewed and approved by Guangdong General Hospital's Ethic Committee, and all participants provided written informed consents. The study will be a prospective, randomized,controlled,single-blind, multi-centre, withdrawal study conducted by Guangdong general hospital, Guangdong Academy of Medical Sciences.there will be two phases, phase 1, Screening and enrolling 112 HBV-GN patients about one year,and phase 2, ongoing follow-up for 24 weeks.The data of all patients will be recorded in the HBV-GN electronic database.Before the randomisation, All patients will receive entecavir routine antiviral therapy for two weeks.And then they will be randomized to two different group,the treatment group: Tacrolimus combined with entecavir antiviral therapy,the control group: The Tacrolimus placebo and entecavir antiviral therapy. The Tacrolimus target trough concentration was 5-10 ng/mL during the therapy. The primary outcome variables were the number of patients who reached complete or partial remission (CR or PR) after the 25 week-treatment. CR was deﬁned as <0.3 g/24 h proteinuria (UPCR<300mg/g.cr) or lower plus stable renal function (eGFR>50 ml/min/1.73 m2) and PR as proteinuria 0.3-3.0 g/24 h (UPCR 300-3000mg/g.cr) and 50% lower than baseline proteinuria plus stable renal function. Secondary outcome variables: 1) The number of patients who reached complete or partial remission (CR or PR) after the 13 week-treatment. 2) Serum creatinine (SCr) increased 2 times the baseline levels or 50% lower than the baseline eGFR(according to chronic kidney disease-EPI (CKD-EPI) )after the 25 week-treatment. 3)Serum HBV DNA was undetectable(HBV DNA<500copies/ml) at the end of 25 week-treatment. 4) The number of patients who present acute kidney injury at the end of 25 week-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 18 and 65 years with HBV-GN;
* All HBV-GN cases with biopsy-proven;
* Evidence of chronic HBV infection based on the presence of HBsAg, HBeAg or HBV DNA in the serum;(HBsAg, HBeAg was positive, HBV DNA ≥10*3 IU/ml). Chronic HBV infection lasted for six months, and all patients did not receive the antiviral therapy in the past six months;
* Proteinuria more than 3.0g/24h, UPCR>3000mg/g.cr, the result will be proofed by at least two tests;
* No glucocorticoid and immunosuppressive treatment within the previous 2 weeks.

Exclusion Criteria:

* The diagnosis of idiopathic membranous nephropathy(MN), systemic lupus erythematosus, malignancy, diabetes mellitus, severe infections or any other systemic disease known to be associated with secondary MN;
* eGFR<30ml/min.1.73m*2;
* Renal pathology showed that Tubular atrophy or Interstitial fibrosis was more than 50%;
* The participant is allergy to tacrolimus, entecavir;
* History of diabetes mellitus;
* History of severe heart disease or cerebrovascular diseases;
* Other active infection such as cytomegalovirus (CMV),Tuberculosis,Hepatitis A virus (HAV),Hepatitis C virus (HCV),Hepatitis D virus (HDV); Innate or acquired immunodeficiency; liver cirrhosis, liver malignment tumor;
* Pregnant, trying to become pregnant or breast feeding;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Remission rate of proteinuria | 25 weeks
  the number of patients who reached complete or partial remission (CR or PR) after the 25 week-treatment. CR was deﬁned as <0.3 g/24 h proteinuria (UPCR<300mg/g.cr) or lower plus stable renal function (eGFR>50 ml/min/1.73 m2) and PR as proteinuria 0.3-3.0 g/24 h (UPCR 300-3000mg/g.cr) and 50% lower than baseline proteinuria plus stable renal function.

SECONDARY OUTCOMES:
Remission rate of proteinuria | 13 weeks
  The number of patients who reached complete or partial remission (CR or PR) after the 13 week-treatment.
The change of Scr | 25 weeks
  SCr increased 2 times the baseline levels or 50% lower than the baseline eGFR(according to CKD-EPI)
Serum HBV DNA | 25 weeks
  Serum HBV DNA was undetectable(HBV DNA<500copies/ml) at the end of 25 week-treatment.
The rate of acute kidney injury | 25 weeks
  The number of patients who present acute kidney injury at the end of 25 week-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Ye, PHD, Study Chair — Guangdong General Hospital, Guangdong Academy of Medical Sciences; Lifen Wang, PHD, Principal Investigator — Guangdong General Hospital, Guangdong Academy of Medical Sciences; Lixia Xu, PHD, Principal Investigator — Guangdong General Hospital, Guangdong Academy of Medical Sciences; Xinling Liang, PHD, Principal Investigator — Guangdong General Hospital, Guangdong Academy of Medical Sciences; Wei Shi, PHD, Study Director — Guangdong General Hospital, Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lai KN, Li PK, Lui SF, Au TC, Tam JS, Tong KL, Lai FM. Membranous nephropathy related to hepatitis B virus in adults. N Engl J Med. 1991 May 23;324(21):1457-63. doi: 10.1056/NEJM199105233242103. PMID 2023605
- [Result] Venkataseshan VS, Lieberman K, Kim DU, Thung SN, Dikman S, D'Agati V, Susin M, Valderrama E, Gauthier B, Prakash A, et al. Hepatitis-B-associated glomerulonephritis: pathology, pathogenesis, and clinical course. Medicine (Baltimore). 1990 Jul;69(4):200-16. PMID 2142748
- [Result] Elewa U, Sandri AM, Kim WR, Fervenza FC. Treatment of hepatitis B virus-associated nephropathy. Nephron Clin Pract. 2011;119(1):c41-9; discussion c49. doi: 10.1159/000324652. Epub 2011 Jun 15. PMID 21677438
- [Result] Tang S, Lai FM, Lui YH, Tang CS, Kung NN, Ho YW, Chan KW, Leung JC, Lai KN. Lamivudine in hepatitis B-associated membranous nephropathy. Kidney Int. 2005 Oct;68(4):1750-8. doi: 10.1111/j.1523-1755.2005.00591.x. PMID 16164651
- [Result] Igarashi T, Shimizu A, Igarashi T, Hanaoka K, Yoshizaki K, Shigemori T, Shimizu S, Komeichi H, Itoh Y. Seroconversion of hepatitis B envelope antigen by entecavir in a child with hepatitis B virus-related membranous nephropathy. J Nippon Med Sch. 2013;80(5):387-95. doi: 10.1272/jnms.80.387. PMID 24189358
- [Result] Zheng XY, Wei RB, Tang L, Li P, Zheng XD. Meta-analysis of combined therapy for adult hepatitis B virus-associated glomerulonephritis. World J Gastroenterol. 2012 Feb 28;18(8):821-32. doi: 10.3748/wjg.v18.i8.821. PMID 22371643
- [Result] Yan H, Zhong G, Xu G, He W, Jing Z, Gao Z, Huang Y, Qi Y, Peng B, Wang H, Fu L, Song M, Chen P, Gao W, Ren B, Sun Y, Cai T, Feng X, Sui J, Li W. Sodium taurocholate cotransporting polypeptide is a functional receptor for human hepatitis B and D virus. Elife. 2012 Nov 13;1:e00049. doi: 10.7554/eLife.00049. PMID 23150796
- [Result] Watashi K, Sluder A, Daito T, Matsunaga S, Ryo A, Nagamori S, Iwamoto M, Nakajima S, Tsukuda S, Borroto-Esoda K, Sugiyama M, Tanaka Y, Kanai Y, Kusuhara H, Mizokami M, Wakita T. Cyclosporin A and its analogs inhibit hepatitis B virus entry into cultured hepatocytes through targeting a membrane transporter, sodium taurocholate cotransporting polypeptide (NTCP). Hepatology. 2014 May;59(5):1726-37. doi: 10.1002/hep.26982. Epub 2014 Apr 1. PMID 24375637
- [Result] Chen M, Li H, Li XY, Lu FM, Ni ZH, Xu FF, Li XW, Chen JH, Wang HY; Chinese Nephropathy Membranous Study Group. Tacrolimus combined with corticosteroids in treatment of nephrotic idiopathic membranous nephropathy: a multicenter randomized controlled trial. Am J Med Sci. 2010 Mar;339(3):233-8. doi: 10.1097/MAJ.0b013e3181ca3a7d. PMID 20220333
- [Result] Chen Y, Schieppati A, Cai G, Chen X, Zamora J, Giuliano GA, Braun N, Perna A. Immunosuppression for membranous nephropathy: a systematic review and meta-analysis of 36 clinical trials. Clin J Am Soc Nephrol. 2013 May;8(5):787-96. doi: 10.2215/CJN.07570712. Epub 2013 Feb 28. PMID 23449768
- [Result] Xu J, Zhang W, Xu Y, Shen P, Ren H, Wang W, Li X, Pan X, Chen N. Tacrolimus combined with corticosteroids in idiopathic membranous nephropathy: a randomized, prospective, controlled trial. Contrib Nephrol. 2013;181:152-62. doi: 10.1159/000348475. Epub 2013 May 8. PMID 23689577
- [Result] Praga M, Barrio V, Juarez GF, Luno J; Grupo Espanol de Estudio de la Nefropatia Membranosa. Tacrolimus monotherapy in membranous nephropathy: a randomized controlled trial. Kidney Int. 2007 May;71(9):924-30. doi: 10.1038/sj.ki.5002215. Epub 2007 Mar 21. PMID 17377504
- [Derived] Xie XF, Xie BY, Zhang WH, Hou JH, Liu DL, Zhang L, Xu LX, Li ZL, Li RZ, Ye ZM. The efficacy and safety of tacrolimus and entecavir combination therapy in the treatment of hepatitis B virus-associated glomerulonephritis: a multi-center, placebo controlled, and single-blind randomized trial. Ann Palliat Med. 2022 May;11(5):1762-1773. doi: 10.21037/apm-22-328. PMID 35672893